CLINICAL TRIAL: NCT07278154
Title: Proprioceptive Neuromuscular Facilitation Versus Music Therapy in Ataxic Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/12/0003; 042111865865 (Other Grant/Funding Number: University of Lahore)
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study will be single and assessor blinded. Participants will be masked about other groups but they will know what treatment they will be receiving or what exercises they will be doing. Principal investigator would also not be masked or blinded because investigator would be applying the techniques on participants of both group. So participant and and principal investigator cannot be blinded. Only assessor will be blinded and he will take outcome measures without knowing the problem and treatment techniques.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (PNF +Conventional physical therapy ) (Experimental): Participants in Group A (PNF Therapy) will receive a structured, minimized treatment plan focused on improving muscle tone, flexibility, and motor function while ensuring the sessions remain tolerable for children with CP. Each session, lasting 20-30 minutes, three times per week, will begin with a 5-minute warm-up, including passive stretching and light joint mobilization. The core intervention will consist of 15 minutes of PNF techniques, such as Rhythmic Initiation, where movements transition from passive to active-assisted, Hold-Relax techniques for reducing spasticity through isometric contractions followed by passive stretching, and Slow Reversals, alternating muscle contractions to improve control. Functional movement patterns with minimal resistance will be incorporated to encourage active participation. The session will conclude with a 5-minute cool-down, focusing on gentle stretching and relaxation techniques to promote comfort and prevent fatigue.
  Interventions: Other: (PNF +Conventional physical therapy ); Other: Music Therapy + Conventional Physical Therapy
- Music Therapy + Conventional Physical Therapy (Experimental): Conversely, participants in Group B (Music Therapy) will engage in 30-minute sessions, three times per week, designed to enhance motor coordination, communication, and emotional well-being through music-based interventions. Each session will start with a 5-10-minute warm-up, incorporating sensory regulation through soft background music, rhythmic swaying, and simple vocal exercises. The 25-minute core intervention will involve Rhythmic Auditory Stimulation (RAS), using rhythmic beats to improve movement control, instrumental play (e.g., drums, xylophone) to enhance upper limb coordination, and movement-to-music activities, such as reaching and stepping in sync with melodies. Additionally, vocal and speech exercises will be incorporated to improve breath control and verbal communication. Sessions will end with a 5-minute cool-down, featuring calming music and gentle tactile stimulation to help the child relax.
  Interventions: Other: (PNF +Conventional physical therapy ); Other: Music Therapy + Conventional Physical Therapy

INTERVENTIONS:
Other: (PNF +Conventional physical therapy ) — Participants in Group A (PNF Therapy) will receive a structured, minimized treatment plan focused on improving muscle tone, flexibility, and motor function while ensuring the sessions remain tolerable for children with CP. Each session, lasting 20-30 minutes, three times per week, will begin with a 5-minute warm-up, including passive stretching and light joint mobilization. The core intervention will consist of 15 minutes of PNF techniques, such as Rhythmic Initiation, where movements transition from passive to active-assisted, Hold-Relax techniques for reducing spasticity through isometric contractions followed by passive stretching, and Slow Reversals, alternating muscle contractions to improve control. Functional movement patterns with minimal resistance will be incorporated to encourage active participation. The session will conclude with a 5-minute cool-down, focusing on gentle stretching and relaxation techniques to promote comfort and prevent fatigue.
Other: Music Therapy + Conventional Physical Therapy — Conversely, participants in Group B (Music Therapy) will engage in 30-minute sessions, three times per week, designed to enhance motor coordination, communication, and emotional well-being through music-based interventions. Each session will start with a 5-10-minute warm-up, incorporating sensory regulation through soft background music, rhythmic swaying, and simple vocal exercises. The 25-minute core intervention will involve Rhythmic Auditory Stimulation (RAS), using rhythmic beats to improve movement control, instrumental play (e.g., drums, xylophone) to enhance upper limb coordination, and movement-to-music activities, such as reaching and stepping in sync with melodies. Additionally, vocal and speech exercises will be incorporated to improve breath control and verbal communication. Sessions will end with a 5-minute cool-down, featuring calming music and gentle tactile stimulation to help the child relax.

SUMMARY:
This study will recruit eligible participants from the Physical Therapy Department of the University of Lahore Teaching Hospital, obtain informed consent, and randomly assign them by lottery into two groups, with the assessor kept blinded. Group A will receive PNF combined with conventional physiotherapy, involving 20-30-minute sessions three times a week, beginning with a warm-up, followed by PNF techniques such as rhythmic initiation, hold-relax, and slow reversals, and ending with a cool-down to enhance muscle tone, flexibility, and motor control. Group B will receive music therapy along with conventional physiotherapy in 30-minute sessions three times a week, incorporating warm-up sensory regulation, rhythmic auditory stimulation, instrument play, movement-to-music activities, and vocal exercises, concluding with calming music for relaxation. The interventions aim to improve motor coordination, communication, and overall functional outcomes in children with cerebral palsy.

DETAILED DESCRIPTION:
Recruitment: Participants will be recruited from Physical Therapy Department of University of Lahore Teaching Hospital.

Screening: All the referred participants will be assessed for the eligibility criteria. Patients fulfilling the eligibility criteria will be asked to sign the consent forms before entering them to the study.

Randomization and Allocation: All the screened and willing participants will be randomly allocated to two groups (Group A: Pnf technique) and (Group B: Music therapy) by lottery method.

Blinding: This study was a single blinded study in which the assessor was kept blinded.

Intervention:

Group A: (PNF +Conventional physical therapy) Participants in Group A (PNF Therapy) will receive a structured, minimized treatment plan focused on improving muscle tone, flexibility, and motor function while ensuring the sessions remain tolerable for children with CP. Each session, lasting 20-30 minutes, three times per week, will begin with a 5-minute warm-up, including passive stretching and light joint mobilization. The core intervention will consist of 15 minutes of PNF techniques, such as Rhythmic Initiation, where movements transition from passive to active-assisted, Hold-Relax techniques for reducing spasticity through isometric contractions followed by passive stretching, and Slow Reversals, alternating muscle contractions to improve control. Functional movement patterns with minimal resistance will be incorporated to encourage active participation. The session will conclude with a 5-minute cool-down, focusing on gentle stretching and relaxation techniques to promote comfort and prevent fatigue.

Group B : (Music Therapy + Conventional Physical Therapy ) Conversely, participants in Group B (Music Therapy) will engage in 30-minute sessions, three times per week, designed to enhance motor coordination, communication, and emotional well-being through music-based interventions. Each session will start with a 5-10-minute warm-up, incorporating sensory regulation through soft background music, rhythmic swaying, and simple vocal exercises. The 25-minute core intervention will involve Rhythmic Auditory Stimulation (RAS), using rhythmic beats to improve movement control, instrumental play (e.g., drums, xylophone) to enhance upper limb coordination, and movement-to-music activities, such as reaching and stepping in sync with melodies. Additionally, vocal and speech exercises will be incorporated to improve breath control and verbal communication. Sessions will end with a 5-minute cool-down, featuring calming music and gentle tactile stimulation to help the child relax. Throughout the intervention, therapists will adjust session intensity based on each child's tolerance, ensuring a supportive and engaging rehabilitation experience.

Outcome Variables:

* Risk of fall: Fall Efficacy Scale
* Coordination: Developmental Coordination Disorder Questionnaire (DCCQ,07)
* Gross motor function: GMFCS scale

  3 sessions per week of 30 minutes will be provided. Data will be assessed by assessor at baseline, at the end of 8th week, 12th week and at the end of 16th week.

ELIGIBILITY:
Inclusion Criteria:

* Children with ataxic CP will be eligible for this study if they are between 6 to 18 years of age.

  * Both genders i.e boys and girls will participate.
  * Children diagnosed with ataxic Cerebral Palsy according to SCPE (Surveillance of Cerebral Palsy in Europe characterized ataxix CP as impairments in balance, coordination, and controlled movements) definition and classification
  * CP children with their gross motor function ranging from level 1-3 on GMFCS (ambulatory ).
  * Evidence of impaired balance or risk of fall
  * Both the caregiver and patients are willing to participate in this study.
  * Consent will be taken from guardians or caregivers.

Exclusion Criteria:

* Patients below or above the age of 6-18.

  * Patients with Down syndrome or psychiatric problems were excluded.
  * Musculoskeletal problems that contraindicates PNF e.g Juvenile Idiopathic Arthritis (in active phase) and osteogenesis imperfecta .
  * Patients with acute and chronic infectious diseases, coagulation diseases, and progressive cerebral diseases such as neoplasms, surgery from the upper and lower extremity in the last 1 year were excluded.
  * Patients with inherited diseases like trisomy 21 syndrome were excluded.
  * Uncontrolled epilepsy or seizures attack.
  * Severe motor impairment (GMFCS level 5).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Fall Efficacy Scale | 12 weeks
  The Fall Efficacy Scale (FES) measures how confident a person feels performing daily activities without falling.It helps clinicians understand fear of falling and plan treatment to improve safety and independence.
Developmental Coordination Disorder Questionnaire (DCDQ-07) | 12 weeks
  The Developmental Coordination Disorder Questionnaire (DCDQ-07) is a parent-report tool used to identify motor coordination difficulties in children aged 5-15.
  It helps screen for Developmental Coordination Disorder by assessing everyday motor skills at home and school.
GMFCS scale | 12 weeks
  It is a five-level scale that describes how children with cerebral palsy move and use mobility aids. It focuses on self-initiated movement-like sitting, standing, and walking-to classify how independently a child functions in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ul Hassan, MS-MSK, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No